CLINICAL TRIAL: NCT01314170
Title: Evaluation of Efficacy and Safety of Susanna Implant in Patients With Refractory Glaucoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adapt Produtos Oftalmológicos Ltda. (Industry)
Responsible Party: PHC - Pharma Consulting, Dr. Dagoberto Brandão
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E01-ADA-VSUS-01-10
Record Dates: First submitted 2010-08-04; First posted 2011-03-14 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Glaucoma
Keywords: Implant, glaucoma, refractory glaucoma.
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Susanna Implant (No Intervention): Patients with refractory glaucoma neovascular type or that failed in trabeculectomy will undergo surgery to place implants Susana.
  Interventions: Device: Susanna Implant

INTERVENTIONS:
Device: Susanna Implant — device
  Other Names: ADA-VSUS-01-10

SUMMARY:
Study clinical multicenter, phase III, open-label, prospective character to evaluate the efficacy and safety Susanna Implant in patients with refractory glaucoma.

DETAILED DESCRIPTION:
Clinical trial multicenter, phase III,open-label, prospective character to evaluate the efficacy and safety of Susanna Implant in patients with refractory glaucoma of both genders, of any race, aged above 18 years and diagnosed with glaucoma refractory.

ELIGIBILITY:
Inclusion Criteria:

Neovascular glaucoma group:

1. Patient with neovascular glaucoma whose intraocular pressures which must be above 21 in at least three measurements, at different times in at least two different days during one month, despite maximum tolerated medical therapy.
2. Visual acuity better than hand movements in the study eye.
3. Patients 18 years or more.
4. Patients with fixed residence in the health district where the surgery will be performed.
5. Patients who fit the term of consent.

Group post-trabeculectomy failure:

1. Patients diagnosed with primary open angle glaucoma, pseudoesfoliação, pigmented or primary angle closure who underwent surgery with trabeculectomy procedure after failure of at least two months of surgery. The pressure must be above 21 in at least three measurements, at different times in at least two different days during one month, despite maximum tolerated medical therapy.
2. Patients diagnosed with primary open angle glaucoma, pseudoesfoliação, pigmented or primary angle closure who underwent surgery with trabeculectomy procedure after failure of at least two months for surgery and who can not afford the expenses of medical treatment. The pressure must be above 21 in at least three measurements, at different times in at least two different days during one month.
3. Visual acuity better than hand movements in the study eye.
4. Patients 18 years or more.
5. Patients with fixed residence in the health district where the surgery will be performed.
6. Patients who fit the term of consent.

Exclusion Criteria:

Group post-trabeculectomy failure:

1. Presence of staphyloma that does not allow the procedure.
2. Presence of history of scleritis
3. Presence of psychiatric disorder that has required hospitalization.
4. Presence of retinal detachment surgery with placement of a buckle or track.
5. Presence of corneal opacity that could prevent the adequate view of the anterior chamber.
6. Presence of shallow anterior chamber that would prevent the placement of the implant.
7. Presence of vitreous in aphakia or anterior chamber.
8. Presence of psychiatric disorder that has required hospitalization.

Neovascular glaucoma group:

1. Presence of staphyloma that does not allow the procedure.
2. Presence of history of scleritis.
3. Presence of corneal opacity that could prevent the adequate view of the anterior chamber.
4. Presence of shallow anterior chamber that would prevent the placement of the implant.
5. Presence of vitreous in aphakia or anterior chamber.
6. Presence of retinal detachment surgery with placement of a buckle or track.
7. Presence of neovascular glaucoma or other secondary glaucoma.
8. Presence of psychiatric disorder that has required hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Study clinical multicenter, phase III, open-label, prospective character to evaluate the efficacy and safety Susanna implant in patients with refractory glaucoma. | 180 days
  Evaluate the effectiveness of implant susanna in patients with refractory glaucoma.

SECONDARY OUTCOMES:
Study clinical multicenter, phase III, open-label, prospective character to evaluate the efficacy and safety Susanna implant in patients with refractory glaucoma. " | 180 days
  Evaluate the safety of implant susanna in patients with refractory glaucoma. i

CONTACTS AND LOCATIONS:
Overall Officials: Remo Susanna, Investigator, Principal Investigator — Hospital das Clínicas de São Paulo; Renato Lisboa, Investigator, Principal Investigator — UNIFESP - Universidade Federal de São Paulo; Cláudia Galvão, Investigator, Principal Investigator — Hospital Universitário Prof. Edgar Santos - BA; Flávia Villas, Investigator, Principal Investigator — - Instituto brasileiro de Oftalmologia e prevenção da cegueira- BA; Fábio Kanadani, Investigator, Principal Investigator — Hospital Universitário São José - Belo Horizonte; Augusto Paranhos, Investigator, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil